## Expanded Preoperative Survey during Perioperative Care to Identify Substance Use in Teenagers and Adolescents – Statistical Analysis Plan

NCT05353036

March 16, 2022

Statistical analysis will be conducted using Python (Python Software Foundation). Chi-squared testing will be used to compare the REDCap patient survey response to the EPIC parental survey data for each substance and to compare categorical demographic data to reports of substance use.